CLINICAL TRIAL: NCT04264767
Title: Characterization of Methylation Patterns in Cancer and Non-Cancer cfDNA, An Observational Multicenter Study
Brief Title: Characterization of Methylation Patterns in Cancer and Non-Cancer cfDNA
Status: Completed | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PNC-RND-UR-001
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Cancer; Solid Tumor; Hematologic Neoplasms
Keywords: Cancer; Methylation; cfDNA; Solid Tumor; Hematologic Neoplasms
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases Group: Peripheral blood collection via routine venipuncture
  Interventions: Procedure: Blood collection
- Control Group: Peripheral blood collection via routine venipuncture
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Peripheral blood collection via routine venipuncture

SUMMARY:
Nucleix EpiCheck® tests analyzes the methylation pattern in a panel of DNA methylation biomarkers and determines whether this pattern is consistent with cancer under test or with non-cancer tissue.

This study is being performed as part of the development process of the Pan Cancer EpiCheck test which includes the identification of different methylation profiles in various cancer types and healthy controls.

DETAILED DESCRIPTION:
The aim of this study is to characterize methylation patterns that will distinguish cancer from normal samples and will be able to recognize the origin of the cancer by collecting cfDNA (circulating free DNA) from blood samples collected from patients with a new diagnosis of cancer and from healthy volunteers who do not have diagnosis or history of cancer. Identifying those methylation patterns may assist in the development of blood test that will be able to detect the presence and the origin of wide range of human cancers

ELIGIBILITY:
Inclusion Criteria - Cases:

1. Age ≥ 22 years
2. Subjects who are willing and able to provide written informed consent.
3. Subjects with confirmed diagnosis of cancer (primary or recurrent) at all stages, however did not yet undergo any surgery, chemotherapy, radiation or any other treatment for this cancerous lesion (including, but not limited to systemic therapies). Recent cancer staging should be within 60 days prior to baseline visit.

Exclusion Criteria - Cases:

1. Known prior diagnosis of cancer except of:

   1. Fully resected non-melanoma skin cancer
   2. History of the original cancer in cases of recurrent disease.
2. Current co-diagnosis of another type of cancer.
3. Currently receiving, or ever received, any of the following therapies to treat their current cancer: surgical management of the cancer beyond that required to establish the cancer diagnosis; local, regional or systemic chemotherapy including chemoembolization; targeted therapy, immunotherapy including cancer vaccines; hormone therapy; or radiation therapy
4. Pregnancy (by self-report)
5. Current febrile illness
6. Acute exacerbation or flare of an inflammatory condition requiring escalation in medical therapy within 14 days prior to blood draw.
7. Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant

Inclusion Criteria - Controls:

1. Age 45 to 80 years
2. Subjects who are willing and able to provide written informed consent

Exclusion Criteria - Controls:

1. Known current or prior diagnosis of cancer except of fully resected non-melanoma skin cancer
2. Currently in work-up due to suspicion of cancer of any kind
3. Oral or IV corticosteroid use in past 14 days prior to blood draw
4. Pregnancy (by self-report)
5. Current febrile illness
6. Acute exacerbation or flare of an inflammatory condition requiring escalation in medical therapy within 14 days prior to blood draw.
7. Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
8. Life expectancy < 24 months

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cases group will include subjects of at least 22 years old that were already diagnosed with cancer but did not yet undergo any surgery, chemotherapy, radiation or any other treatment for this cancer (i.e. treatment naïve subjects). Enrollment for this group will be stratified to enable representation of subjects with multiple tumor histological types, stage and grade.
  The control group will include healthy subjects, 45-80 years old. The subjects in the control group should be without any previous or current diagnosis of cancer except completely resected non-melanoma skin cancer.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
To collect blood and urine samples and clinical data in order to characterize methylation patterns that will discriminate cancer and normal (non-cancer) samples and the origin of cancer | 72 Months
  To collect blood and urine samples and clinical data in order to characterize methylation patterns that will discriminate cancer and normal (non-cancer) samples and the origin of cancer
To develop a molecular blood test that will be able to detect wide range of human cancers based on change in methylation patterns between cancer and normal samples | 72 Months
  To develop a molecular blood test that will be able to detect wide range of human cancers based on change in methylation patterns between cancer and normal samples

CONTACTS AND LOCATIONS:
Overall Officials: Shmulik Adler, Study Director — Nucleix Ltd.
Locations (3):
- United States (2):
  - Los Angeles Hematology Oncology Medical Group - Wilson Terrace, Glendale, California
  - Los Angeles Hematology Oncology Medical Group - Good Samaritan Medical Offices, Los Angeles, California
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. The analysis will be performed by the sponsor